CLINICAL TRIAL: NCT06511856
Title: Observational Study of Shoulder Surgery Using FH ORTHO Medical Devices
Brief Title: FH ORTHO Shoulder Observatory
Status: Recruiting | Type: Observational
Sponsor: FH ORTHO (Industry)
Responsible Party: Sponsor
Other Study IDs: 2020-03
Record Dates: First submitted 2024-07-08; First posted 2024-07-22 (Actual); Last update posted 2024-07-22 (Actual); Status verified 2024-07

CONDITIONS: Trauma; Arthropathy Shoulder
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- FH ORTHO shoulder patients: Patients operated with FH ORTHO shoulder medical devices (arthroplasty and trauma)
  Interventions: Device: ARROW

INTERVENTIONS:
Device: ARROW — Patients included in the study are patients operated with one or more shoulder medical device fabricated by FH ORTHO. Medical devices of interest are CE marked and include ARROW and ARROW prosthesis, Telegraph Evolution humeral nail and STRAPFLEX strapping system.
  Other Names: ARROW II; Telegraph Evolution; STRAPFLEX

SUMMARY:
This study is a real-life observatory designed to collect long-term clinical data on patients who have undergone shoulder joint replacement or repair following shoulder trauma.

In this type of intervention, one or more medical devices distributed by FH ORTHO SAS may be used by surgeons.

This study meets the requirement for post-market clinical follow-up (PMCF) as defined in the European Medical Device Regulation (MDR 2017/745).

It therefore involves collecting in real life, i.e. under the usual conditions of surgery and short and long-term patient follow-up, minimal clinical data that will make it possible to document the continued benefit/risk of the medical devices concerned.

This study is designed as a permanent long-term observatory, of a non-interventional nature, with the objective of having long-term follow-up data (5 to 10 years depending on the devices concerned) for a maximum number of patients included.

ELIGIBILITY:
Inclusion criteria:

1. Any patient undergoing implantation of medical devices distributed by FH ORTHO SAS for shoulder arthroplasty and traumatology, used in accordance with their approved labelling, in one of the centres participating in the Observatory (retrospectively or prospectively)
2. Patient is at least 18 years of age
3. Patient agreeing to participate after having been informed orally and in writing (with written consent if required locally) In some countries, such as France, the patient will have to be socially insured to be included in the study.

Exclusion criteria:

1. Patient unable to participate in the study and/or complete the questionnaires 2. Refusal of patient participation

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any patient considered for implantation or use of medical devices for shoulder arthroplasty and traumatology distributed by FH ORTHO SAS.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2022-09-08 (Actual); Primary Completion 2032-09-08 (Estimated); Study Completion 2035-09-08 (Estimated)

PRIMARY OUTCOMES:
Performance of the medical devices over long term follow-up (maximum10 years) | maximum 10 years
  Functional performance measured by the Constant-Murley score

SECONDARY OUTCOMES:
revision rate medical devices over long term follow-up (maximum10 years) | maximum 10 years

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - Clinique VIA DOMITIA, Lunel
  - Clinique Bizet, Paris
  - Clinique de l'Union, Saint-Jean